CLINICAL TRIAL: NCT00011895
Title: A Phase IV Multicenter Study of the Efficacy and Safety of 48-Week Induction Treatment With TRIZIVIR (Abacavir 300 Mg/Lamivudine 150 Mg/Zidovudine 300 Mg Combination Tablet BID) With Efavirenz (600 Mg QD) Followed by 48-Week Randomized, Open-Label, Maintenance Treatment With TRIZIVIR With or Without Efavirenz in HIV-1 Infected Antiretroviral Therapy Naive Subjects
Brief Title: Safety and Effectiveness of TRIZIVIR (Abacavir/Lamivudine/Zidovudine) With Efavirenz in HIV-Infected Patients Who Have Never Taken Anti-HIV Drugs
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: GlaxoSmithKline (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 308B; ESS40013
Record Dates: First submitted 2001-03-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2002-03

CONDITIONS: HIV Infections
Keywords: HIV-1; Drug Therapy, Combination; Zidovudine; Lamivudine; Drug Combinations; RNA, Viral; Reverse Transcriptase Inhibitors; Anti-HIV Agents; Viral Load; abacavir; efavirenz
MeSH Terms: conditions — HIV Infections | interventions — abacavir; Lamivudine; Zidovudine; efavirenz

INTERVENTIONS:
Drug: Abacavir sulfate, Lamivudine and Zidovudine
Drug: Efavirenz

SUMMARY:
The purpose of this study is to determine the effect of treatment with Trizivir (TZV) plus efavirenz (EFV) or TZV alone on viral load (level of HIV in the blood).

DETAILED DESCRIPTION:
Patients receive TZV plus EFV in the 48-week Induction Phase. Eligible patients, defined as those with plasma HIV-1 RNA under 50 copies/ml, participate in the 48-week Maintenance Phase. Patients are randomized equally to receive either TZV plus EFV or TZV alone.

An immunology substudy will be conducted, including approximately the first 100 patients enrolled who agree to participate.

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible for this study if they:

* Are at least 13 years old.
* Are HIV-positive.
* Have a viral load of at least 5,000 copies/ml.
* Agree to use adequate and reliable methods of birth control. Note: Hormonal birth control is not considered adequate.
* Provide written consent of a parent or guardian, if under 18 years of age.

Exclusion Criteria

Patients will not be eligible for this study if they:

* Have taken nonnucleoside reverse transcriptase inhibitors.
* Have taken other anti-HIV drugs for 2 weeks or more.
* Have an opportunistic (AIDS-related) infection.
* Are pregnant or breast-feeding.
* Have had hepatitis within the past 6 months.
* Are allergic to the study drugs or their ingredients.
* Have a mental, physical, or substance abuse disorder.
* Have a serious medical condition, such as diabetes, congestive heart failure, or other heart disease.
* Have a gastrointestinal disorder that affects drug absorption or makes it difficult to take medication by mouth.
* Have received within 4 weeks before study entry, or may require during the study period, radiation therapy, chemotherapy, or drugs that affect the immune system (such as steroid drugs, interleukins, vaccines, or interferons).
* Have received an HIV vaccine within 3 months before study entry, or are scheduled to receive one during the study period.
* Require foscarnet or other drugs that are shown to be effective against HIV.
* Are taking astemizole, cisapride, midazolam, triazolam, or ergot derivatives.
* Are taking experimental drugs.
* Are unlikely to complete the study or take the drugs.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400
Dates: Start 2001-02

CONTACTS AND LOCATIONS:
Locations (42):
- United States (42):
  - Phoenix Body Positive, Phoenix, Arizona
  - Health for Life Clinic, Little Rock, Arkansas
  - Orange County Ctr for Special Immunology, Fountain Valley, California
  - Pacific Horizons Med Group, San Francisco, California
  - Beacon Clinic / Boulder Community Hosp, Boulder, Colorado
  - Georgetown Univ Med Ctr, Washington D.C., District of Columbia
  - Dupont Circle Physicians Group, Washington D.C., District of Columbia
  - Infectious Disease Consultants, Altamonte Springs, Florida
  - North Broward Hosp District / HIV Clinical Research, Fort Lauderdale, Florida
  - Univ of Miami / Jackson Memorial Hosp, Miami, Florida
  - SBMA Research, Miami Beach, Florida
  - Infectious Disease Specialists of Atlanta, Decatur, Georgia
  - Cook County Gen Hosp / Division of Infect Diseases, Chicago, Illinois
  - Northstar Med Clinic, Chicago, Illinois
  - University of Louisville / ID Division, Louisville, Kentucky
  - HIV Outpatient Clinics / LA State Univ Med Ctr, New Orleans, Louisiana
  - Boston Med Ctr, Boston, Massachusetts
  - Dr Paul Benson, Berkley, Michigan
  - Hennepin County Med Ctr, Minneapolis, Minnesota
  - Regions Hosp / HIV/AIDS Program, Saint Paul, Minnesota
  - CRC of Mississippi, Jackson, Mississippi
  - Wellness Ctr / Las Vegas, Las Vegas, Nevada
  - Hackensack University Medical Center, Hackensack, New Jersey
  - NJCRI, Newark, New Jersey
  - SUNY / Health Sciences Ctr at Brooklyn, Brooklyn, New York
  - Aaron Diamond AIDS Rsch Ctr / Rockefeller Univ, New York, New York
  - ID Consultants, Charlotte, North Carolina
  - East Carolina Univ School of Medicine, Greenville, North Carolina
  - Summa Health System, Akron, Ohio
  - Univ of Oklahoma Infectious Disease Institute, Oklahoma City, Oklahoma
  - Associates in Med and Mental Health, Tulsa, Oklahoma
  - Univ of Tennessee Med Ctr at Knoxville, Knoxville, Tennessee
  - Texas Tech Health Sciences Ctr, El Paso, Texas
  - AIDS Outreach Center, Fort Worth, Texas
  - Metroplex Infectious Disease, Fort Worth, Texas
  - Tarrant County Infectious Diseases Associates, Fort Worth, Texas
  - Therapeutic Concepts, Houston, Texas
  - Diversified Med Practices, PA, Houston, Texas
  - Infectious Diseases Associates of Houston, Houston, Texas
  - Infectious Disease Physicians Inc, Annandale, Virginia
  - Infectious Disease Consultants, Fairfax, Virginia
  - Swedish Med Ctr, Seattle, Washington